CLINICAL TRIAL: NCT01905579
Title: Correlation Between Aqueous Protein Level and Clinical Grading of Flare and Flaremetry.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Principal Investigator, Samir S. Shoughy, MD, FRCS (Glasg.), Ophthalmologist, The Eye Center and The Eye Foundation for Research in Ophthalmology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TEC 123; TEC 2012-003 (Other: THE EYE CENTER)
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Uveitis
Keywords: flaremetry; aqueous proteins; clinical grading; Compare flaremetry readings with the protein content of the aqueous; Compare flaremetry readings with clinical grading of flare
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with uveitis (Experimental): Paracentesis of the anterior chamber in Paients with uveitis undergoing cataract surgery
  Interventions: Procedure: Paracentesis of the anterior chamber
- patients without uveitis (Experimental): Paracentesis of the anterior chamber in patients without uveitis undergoing routine cataract surgery
  Interventions: Procedure: Paracentesis of the anterior chamber

INTERVENTIONS:
Procedure: Paracentesis of the anterior chamber — Aqueous humor parenthesis for quantitative protein analysis in patients with and without uveitis.

SUMMARY:
The purpose of this study is to compare flaremetry readings with the protein content of the aqueous humor and the clinical grading of flare.

DETAILED DESCRIPTION:
A total of 20 patients will be included. 10 patients with uveitis and 10 control patients scheduled for phacoemulsification. Each patient will undego complete ophthalmic examination and clinical biomicroscopic grading of the anterior chamber flare applying the SUN working group grading system. Aqueous specimens will be obtained by anterior chamber paracentesis for protein analysis. Each Patient will undego paracentesis and 0.2 ml of aqueous will be obtained. The aqueous sample will be stored at -70°C until the time of analysis for protein content. Objective assessment of flare will be done.

ELIGIBILITY:
Inclusion Criteria:

* 10 patients with uveitis with cataract
* 10 patients without uveitis with cataract
* Inactive inflammation for at least 3 months

Exclusion Criteria:

* Infectious uveitis
* endophthalmitis
* cases with corneal scar

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
compare flaremetry readings with the protein content of the aqueous humor | one month
  Compare flaremetry readings with the protein content of the aqueous and the clinical grading.

CONTACTS AND LOCATIONS:
Overall Officials: Samir S Shoughy, Principal Investigator — THE EYE CENTER
Locations (1):
- The Eye Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Shoughy SS, Elkum N, Tabbara KF. Aqueous protein level and flare grading. Acta Ophthalmol. 2015 Mar;93(2):e173-4. doi: 10.1111/aos.12522. Epub 2014 Aug 31. No abstract available. PMID 25175512